CLINICAL TRIAL: NCT03840863
Title: Effects of Chronic Energy Drink Consumption on Cardiometabolic Endpoints
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Pacific (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19-02
Record Dates: First submitted 2019-01-11; First posted 2019-02-15 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Cardiovascular Diseases
Keywords: Energy Drink; Blood Pressure; Arrhythmia
MeSH Terms: conditions — Cardiovascular Diseases; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Commercially-Available Energy drink (Experimental): Healthy volunteers willing to consume two cans of energy drinks (16 oz./can) daily for 4 weeks
  Interventions: Dietary Supplement: Commercially-Available Energy Drink

INTERVENTIONS:
Dietary Supplement: Commercially-Available Energy Drink — Participant will consume 2 cans of an energy drink (16 oz./can) per day. One in the morning and one in the afternoon.

SUMMARY:
Many people use energy drinks (EDs) regularly, but the overall health concerns are still unknown. There are many energy drink products that contain a mixture of caffeine and other energy-boosting ingredients and supplements which can affect parameters related to the heart, blood pressure and blood glucose. Several previous studies have shown that energy drinks may affect heart rhythm and blood pressure significantly. As energy drinks are sugar-sweetened beverages, long-term use may also affect the body's metabolism, including cholesterol, blood sugars, and weight.

The purpose of this study is to learn if drinking energy drinks everyday may affect a person's cardiometabolic health.

DETAILED DESCRIPTION:
The popularity of energy drinks (EDs) have increased over the last few decades due to their purported benefits as mental and physical performance enhancements. While caffeine is a major ingredient in most EDs (ranging from 80 mg to 500 mg per drink), they may also contain various supplements, such as guarana, taurine, ginseng, B vitamins, gluconolactone, yohimbe, carnitine, and bitter orange, as well as high amount of sugar (ranging from 25-50 grams). The United States Food and Drug Administration (FDA) has cited that a daily intake of 400 mg caffeine (approximately 4-5 cups of coffee) in adults is generally safe and not associated with dangerous, negative effects. The Substance Abuse and Mental Health Services Administration reported a doubling of emergency department visits involving EDs from 10,068 visits in 2007 to 20,783 visits in 2011. Commonly reported adverse reactions include insomnia, nervousness, headache, tachycardia, and seizures. Currently, the health effects of long-term ED use remain unknown.

This study is a proof-of-concept, prospective trial that aims to evaluate the effects of chronic ED consumption on cardiometabolic parameters in a healthy population. Subjects will consume two cans (16 oz.) of an energy drink daily for 4 weeks. The study will assess any changes in blood pressure (BP), electrocardiographic (ECG) parameters, blood glucose, cholesterol, weight, body mass index (BMI), and body fat composition before and after consuming EDs for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 - 40 years
* Participants willing to adhere to study drink schedule (28 days)

Exclusion Criteria:

* Naïve caffeine consumers (< 2 cups of coffee [or equivalent caffeine intake] per week)
* Chronic medical conditions including cardiovascular disease (known history of cardiac arrhythmias, family history of premature sudden cardiac death before age 60, cardiomyopathy, atherosclerosis), smoking, renal or hepatic dysfunction
* Prolonged corrected QT (QTc) interval
* History of substance abuse, including alcohol
* Concurrent use of prescription drugs or over-the-counter products that may interact with study drinks (with the exception of oral contraceptives that have been used for over 1 month)
* Baseline Blood Pressure greater than 140/90 mmHg
* Baseline fasting blood glucose greater than 126 mg/dL or random blood glucose greater than 200 mg/dL
* Females only: pregnancy or lactation, or planning to get pregnant within next 28 days

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure before and 1 hour after energy drink consumption | 1 hour
  Measuring acute changes in peripheral systolic blood pressure before and 1 hour after energy drink consumption
Change in blood pressure before and after 4 weeks of energy drink consumption | 4 weeks
  Measuring chronic changes in peripheral systolic blood pressure before and 4 weeks after energy drink consumption

SECONDARY OUTCOMES:
Change in QTc Interval before and after 1 hour of energy drink consumption | 1 hour
  Measuring change in QTc interval via electrocardiogram before and after 1 hour of energy drink consumption
Change in QTc Interval before and after 4 weeks of energy drink consumption | 4 weeks
  Measuring change in QTc interval via electrocardiogram before and after 4 weeks of energy drink consumption
Change in fasting blood glucose before and after 4 weeks of energy drink consumption | 4 weeks
  Measuring the change in fasting blood glucose before and after 4 weeks of energy drink consumption
Change in fasting lipid panel parameters before and after 4 weeks of energy drink consumption | 4 weeks
  Measuring the changes in total cholesterol (TC), high-density lipoprotein (HDL), triglyceride (TG), and calculated low-density lipoprotein (LDL-C) levels before and after 4 weeks of energy drink consumption
Change in Body Mass Index before and after 4 weeks of energy drink consumption | 4 weeks
  Measuring the change in Body Mass Index (BMI) before and after 4 weeks of energy drink consumption
Change in Body Fat Analysis before and after 4 weeks of energy drink consumption | 4 weeks
  Measuring the changes in Body Fat Analysis before and after 4 weeks of energy drink consumption, including percentage of body fat, fat mass, muscle mass, and fat in trunk
Change in Serum Creatinine before and after 4 weeks of energy drink consumption | 4 weeks
  Measuring the change in Serum Creatinine before and after 4 weeks of energy drink consumption

CONTACTS AND LOCATIONS:
Overall Officials: May Chen, PharmD, Principal Investigator — University of the Pacific
Locations (1):
- University of the Pacific, Stockton, California, United States

IPD SHARING:
Plan to Share IPD: No